CLINICAL TRIAL: NCT00502190
Title: Evaluation Of Pessaries In Twin Pregnancies With A Short Cervix (25 mm) Between 20-28 WG
Brief Title: Evaluation Of Pessaries In Twin Pregnancies With A Short Cervix (25 mm) Between 20-28 WG (EPEGE)
Acronym: EPEGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P050322
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2007-04

CONDITIONS: Twin Pregnancy
Keywords: pessary; extending pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Silicon ring positioned in the vagina, around the cervix
  Interventions: Device: Silicon ring positioned in the vagina, around the cervix
- 2 (Experimental): Silicon ring positioned in the vagina, around the cervix
  Interventions: Device: Silicon ring positioned in the vagina, around the cervix

INTERVENTIONS:
Device: Silicon ring positioned in the vagina, around the cervix — Silicon ring positioned in the vagina, around the cervix

SUMMARY:
Randomized, opened multicentric study evaluating the Effectiveness of Pessary in the patients with a Gemellary pregnancy and a collar runs between 20 and 28 weeks of amenorrhoea

DETAILED DESCRIPTION:
Randomized, opened multicentric study evaluating the Effectiveness of Pessary in the patients with a Gemellary pregnancy and a collar runs between 20 and 28 weeks of amenorrhoea To show that the use of pessary makes it possible to lengthen the duration of the pregnancy of at least 10 days in patients with a twin pregnancy and a uterine collar length < = 25 mm measured by echography between 20 and 28 SA compared to the group controls.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years (legal majority in France)
* Inclusion pessary positioning before 28 WG
* Twin pregnancies, mono or dichorionic, diamniotic
* Transvaginal cervical length ( 25mm between 20 et 28 WG
* Intact membranes
* No signs of infection (negative urine culture, CRP <10mg/l , blood white cell count <15000/ml)
* Patient accepting follow-up
* Covered by health insurance for France

Exclusion Criteria:

* Cerclage

  * No more cervix
  * Chorioamnionitis
  * Abnormal CTG
  * Placenta praevia
  * Abruptio
  * Bleeding
  * PROM
  * Singleton or multiple >2
  * Monochorionic monoamniotic twin pregnancy
  * IUGR
  * Preeclampsia or other PIH
  * TTTS
  * Uncontrolled diabetes
  * Other maternal of fetal pathology responsible for preterm deliveries
  * Patient included in other therapeutic trials
  * Patient without legal freedom to consent
  * Homeless or no fixed address

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Demonstrate the profit of 10 days in the pessary group compared to control. | at least 10 days
  Demonstrate the profit of 10 days in the pessary group compared to control

SECONDARY OUTCOMES:
To evaluate and compare the frequency of the childbirth < 34 SA | before 34 weeks
Deliveries (<34WG) | 34 weeks
  Deliveries (<34WG)
Evaluate the rate of side effects of pessaries | during the pessaries
  Evaluate the rate of side effects of pessaries
Neonatal outcome | before 28 weeks
  Neonatal outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jacky NIZARD, CCA, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital POISSY-ST GERMAIN EN LAYE, Poissy, France